CLINICAL TRIAL: NCT01823003
Title: Risk Adapted Free Flattering Filter Based Stereotactic Ablative Radiotherapy (Sabr) in Stage i Nsclc and Lung Metastases
Brief Title: Risk Adapted SABR(SABR) in Stage I NSCLC And Lung Metastases
Acronym: sbrtlungfff
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sbrt_lung_fff2012
Record Dates: First submitted 2013-03-25; First posted 2013-04-04 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis
Keywords: Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Radiosurgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A. 34 Gy in a single fraction (Experimental): 34 Gy by single fraction Risk-adapted radiation dose.
  Interventions: Radiation: 34 Gy in a single fraction
- B. 54Gy (18Gy/fr. x 3 fractions) (Experimental): 54Gy administered in 3 fraction of 18 Gy, risk adapted radiation dose
  Interventions: Radiation: 54Gy 18Gy/fr. x 3 fractions
- C. 50Gy (12 x 5 fr.s) (Experimental): 54Gy administered in 5 fraction of 12 Gy, risk adapted radiation dose
  Interventions: Radiation: 60Gy (12 x 5 fr.s)
- D. 60Gy (7.5Gy x 8fr.) (Experimental): 60 Gy administered in 8 fraction of 7.5 Gy, risk adapted radiation dose
  Interventions: Radiation: 60Gy (7.5Gy x 8fr.)

INTERVENTIONS:
Radiation: 34 Gy in a single fraction — 34 Gy in a single fraction in case of Distance to chest wall > 1 cm, tumour size < 2 cm and distance to the main bronchus > 2 cm. STEREOTACTIC ABLATIVE RADIOTHERAPY (SABR) will be administered with volumetric modulated arcs, with photon beam energy of 6-10 MV. The number of arcs and their ballistic is left undefined in order to allow for optimization of the dose distribution. Bolus is not allowed.
  Arms: A. 34 Gy in a single fraction
Radiation: 54Gy 18Gy/fr. x 3 fractions — 54Gy administered in 3 fractions of 18Gy in case of distance to chest wall > 1 cm, tumour size between 2 and 5 cm and distance to the main bronchus > 2 cm. STEREOTACTIC ABLATIVE RADIOTHERAPY (SABR)will be administered with volumetric modulated arcs, with photon beam energy of 6-10 MV. The number of arcs and their ballistic is left undefined in order to allow for optimization of the dose distribution. Bolus is not allowed.
  Arms: B. 54Gy (18Gy/fr. x 3 fractions)
Radiation: 60Gy (12 x 5 fr.s) — 50Gy administered in 5 fractions of 12 Gy for Peripheral Nodes in case of distance to chest wall < 1 cm, tumour size < 5 cm and distance to main bronchus > 2 cm. STEREOTACTIC ABLATIVE RADIOTHERAPY (SABR) will be administered with volumetric modulated arcs, with photon beam energy of 6-10 MV. The number of arcs and their ballistic is left undefined in order to allow for optimization of the dose distribution. Bolus is not allowed.
  Arms: C. 50Gy (12 x 5 fr.s)
Radiation: 60Gy (7.5Gy x 8fr.) — 60 Gy administered in 8 fractions of 7.5 Gy for mediastinal nodes in case of tumour size < 5 cm and distance to the main bronchus < 2 cm. STEREOTACTIC ABLATIVE RADIOTHERAPY (SABR)will be administered with volumetric modulated arcs, with photon beam energy of 6-10 MV. The number of arcs and their ballistic is left undefined in order to allow for optimization of the dose distribution. Bolus is not allowed.
  Arms: D. 60Gy (7.5Gy x 8fr.)

SUMMARY:
This study is designed to evaluate the safety of Stereotactic Ablative Radiotherapy (SBRT) in selected patients with stage I Non Small Cell Lung Cancer (NSCLC) or metastatic lung cancer to demonstrate the feasibility and risks of using an ablative dose-adapted scheme with FFF beams. Other aims are To evaluate the incidence of acute and late complications; To evaluate tumour response to local radiation therapy by means of CT, PET/TC and MRI and To evaluate the impact of local therapy on overall and disease-free survival.

DETAILED DESCRIPTION:
The intervention (dose and fractions) depends on topographical parameters: lung disease (primary, peripheral nodes or mediastinal nodes), distance to chest wall, tumour size and distance to main bronchus.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed primary lung cancer or lung metastasis from another primary tumour or positive PET/CT suggestive for primary tumour(SUV MAX> 4).
* Tumour size < 5 cm in diameter prior to treatment.
* Medically inoperable patients as determined by the multidisciplinary thoracic tumour board, or medically operable patients who refuse surgery.
* Life expectancy of >12 months.
* Criterion for medical inoperability include:

Overall clinical assessment at the UCLA thoracic tumour board. Reduced Pulmonary Function (FEV1, DLCO, etc) based on one major or two minor criterion as described below: Minor Criteria: Age > 75, FEV1 51- 60% predicted, or FEV1 1-1.2L, DLCO 51%-60% predicted, pulmonary hypertension, poor left ventricular function (EF < 40% or less), resting or exercise arterial pO2 < 55 mmHg, and pCO2 > 45 mmHg.

* Age > 18 years.
* KPS > 70.
* Barthel score >40
* Baseline computed tomography scans of the chest, pulmonary test function, and positron emission tomography no more than 2 months before treatment.
* If a woman is of childbearing potential, a negative urine or serum pregnancy test must be documented.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior thoracic radiation treatment wich dose contribution can be expected in the new SBRT plan.
* More than two lesions per lobe.
* Active infections requiring systemic antibiotics.
* Age <18 years old.
* KPs < 70.
* Barthel Total Score < 40.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2012-06; Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
probability of not suffering a grade 3 or higher toxicity | one year
  Patients will be follow-up during one year. If patient suffered any toxicity grade 3 or higher during this period it will be classified as having toxicity. Otherwise patient will be classified as not having toxicity.

SECONDARY OUTCOMES:
Tumour response | One year
  To evaluate tumour response attending histology with local radiation using imaging such as CT and PET/CT.
Incidence of acute and late toxicities | One year
  To evaluate the frequency of acute and late toxicities.
Overall survival | One year
  To evaluate the impact of local therapy on overall survival.
Disease-free survival | One year
  To evaluate the impact of local therapy on disease-free survival.
Effect in brochopulmonary (COPD) disease. | One year
  To evaluate the impact of local therapy on bronchopulmonary (COPD) disease.
Feasibility | One year
  To evaluate the feasibility of this technique in terms of technical complications.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Navarro-Martin, md, Principal Investigator — Institut Català d'Oncologia L'Hospitalet
Locations (1):
- Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Barcelona, Spain